CLINICAL TRIAL: NCT00318474
Title: A Randomized Controlled Trial of Mycophenolate Mofetil in Patients With IgA Nephropathy
Brief Title: Mycophenolate Mofetil (MMF) in Patients With IgA Nephropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommended stopping the trial because of lack of effect.
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04PE116; IND #48,977 (Other: Food and Drug Administration); Canadian Control #076948 (Other: Bureau of Pharmaceutical Assessment - Canada)
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: IgA Nephropathy
Keywords: Proteinuria; Immunoglobulin A
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Mycophenolic Acid; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil (MMF) (Active Comparator): Dose is based on body size (between 25mg/kg/day and 36mg/kg/day with a maximum dose 1gm BID; initial dose to be used in the first 2 weeks of therapy will be approximately 1/2-2/3 of the full dose). Route of administration is oral. Frequency is daily. MMF will be administered up to 12 months.
  Interventions: Drug: Mycophenolate Mofetil (MMF); Drug: ACEi; Drug: FOS
- MMF Placebo (Placebo Comparator): Subjects receive MMF placebo.
  Interventions: Drug: MMF Placebo; Drug: ACEi; Drug: FOS

INTERVENTIONS:
Drug: Mycophenolate Mofetil (MMF) — Oral administration of MMF; dose based on body size (between 25mg/kg/day and 36ng/kg/day); maximum dose 1gm BID.
  Other Names: CellCept
  Arms: Mycophenolate Mofetil (MMF)
Drug: MMF Placebo — Placebo only, oral administration
  Arms: MMF Placebo
Drug: ACEi — Administer same as pre-treatment regimen.
  Other Names: angiotensin converting enzyme inhibitors
Drug: FOS — Administer same as pre-treatment regimen
  Other Names: fish oil supplement

SUMMARY:
IgA nephropathy (IgAN) is the most common type of glomerulonephritis worldwide. 15-40% of individuals diagnosed with IgAN, including children, will eventually progress to chronic renal insufficiency (CRI) and end stage renal disease (ESRD). The study is to evaluate the safety and benefits of MMF in patients with IgAN who have been pre-treated (and continue to be treated) with angiotensin converting enzyme inhibitors (ACEi) and fish oil supplements (FOS).

DETAILED DESCRIPTION:
A multi-center, randomized, controlled clinical trial to test the hypothesis that treatment with mycophenolate mofetil (MMF) will lead to significant and sustained improvement in proteinuria in patients with IgA Nephropathy who have been pre-treated (and continue to be treated) with ACEi and FOS compared to a placebo control group of patients receiving comparable doses of ACEi and FOS without MMF. Data for this outcome will be examined every six months and at the end of 2 years of study. Comparisons will be made between the two treatment groups for change from entry level in urine protein to creatinine (UPr/Cr) ratio, 24-hour urine protein excretion rate and estimated glomerular filtration rate (GFR).

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 7-70 years old
* Renal biopsy, diagnostic for IgA nephropathy
* Must be able to take oral medication

Exclusion Criteria:

* Clinical and histologic evidence of systemic lupus erythematosus
* Well-documented history of Henoch-Schonlein purpura.
* Clinical evidence of cirrhosis or chronic liver disease
* Abnormal laboratory values at the time of study entry
* Estimated GFR outside of protocol defined limits
* History of significant gastrointestinal disorder
* Active systemic infection or history of serious infection within one month of entry or known infection with HIV, hepatitis B, or hepatitis C.
* Other major organ system disease or malignancy
* Current or prior treatment with MMF or azathioprine

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2002-01; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Hogg, M.D., Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 184 subjects were enrolled. 146 subjects completed entry evaluation. 97 subjects fulfilled entry criteria and were started on 3 month course of Omacor and lisinopril. 94 subjects completed the 3 months of treatment.
Pre-assignment Details: After the 3 months, 58 subjects fulfilled criteria for going into the MMF vs. placebo phase. Six of the 58 subjects were not randomized because the External Advisory Committee/Data Safety Monitoring Board recommended stopping the trial because of lack of effect.
Groups:
- Mycophenolate Mofetil (MMF): Subjects receive angiotensin-converting enzyme inhibitors (ACEi), fish oil supplements (FOS), and MMF. Dose is based on body size (between 25mg/kg/day and 36mg/kg/day with a maximum dose 1gm BID; initial dose to be used in the first 2 weeks of therapy will be approximately 1/2-2/3 of the full dose). Route of administration is oral. Frequency is daily. MMF will be administered up to 12 months.
  Mycophenolate Mofetil (MMF)
- Placebo: Subjects receive ACEi and FOS and placebo.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF) | Placebo
Started | 25 | 27
Completed | 7 | 10
Not Completed | 18 | 17
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Fall in GFR | 3 | 3
Not completed — Post-therapy hyperflycemia | 0 | 1
Not completed — Trial terminated | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Mycophenolate Mofetil (MMF): Subjects receive ACEi, FOS, and MMF. Dose is based on body size (between 25mg/kg/day and 36mg/kg/day with a maximum dose 1gm BID; initial dose to be used in the first 2 weeks of therapy will be approximately 1/2-2/3 of the full dose). Route of administration is oral. Frequency is daily. MMF will be administered up to 12 months.
  Mycophenolate Mofetil (MMF)
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil (MMF) | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (11.7) | 32.2 (13.2) | 32.0 (12.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 14 | 18 | 32
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42
  Canada | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria - Uprotein/Creatinine Ratio
Description: Urine protein/creatinine ratio after 6 months treatment with MMF or placebo.
Time Frame: Plan was to measure uprotein/creatinine ratio for 12 months on MMF or placebo, and then 12 months post-treatment. Data given after 6 months MMF/placebo.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mycophenolate Mofetil (MMF) | Placebo
Number analyzed (Participants) | 25 | 27
ratio | 1.40 (0.72) | 1.58 (1.07)

2. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (GFR) to Less Than 60% of the Baseline Level
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The trial design is 13 visits over 27 months.
Description: Adverse events assessed at each encounter with subject.
Arm/Group | Mycophenolate Mofetil (MMF) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/27
Other Adverse Events (participants affected / at risk) | 25/25 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (MMF) (N=25) | Placebo (N=27)
melanoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
trauma (General disorders) | 1 (1) | 0 (0) — motor vehicle accident (mva)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil (MMF) (N=25) | Placebo (N=27)
backache (Musculoskeletal and connective tissue disorders) | 6 | 6
common cold (Respiratory, thoracic and mediastinal disorders) | 5 | 7
coughing (Respiratory, thoracic and mediastinal disorders) | 9 | 9
diarrhea (Gastrointestinal disorders) | 4 | 6
edema (General disorders) | 5 | 3
heartburn (Gastrointestinal disorders) | 5 | 2
nausea (Gastrointestinal disorders) | 8 | 4
sore throat (Infections and infestations) | 1 | 7
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No